CLINICAL TRIAL: NCT05035771
Title: A Safety and Feasibility Study of Intraprocedural Physiology Measurements During Peripheral Endovascular Treatment
Brief Title: The IMPACT PAD Study
Acronym: IMPACT PAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Essex CTC IMPACT PAD
Record Dates: First submitted 2021-06-21; First posted 2021-09-05 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pressure wire measurements (Experimental)
  Interventions: Device: Pressure wire measurement in peripheral vascular disease

INTERVENTIONS:
Device: Pressure wire measurement in peripheral vascular disease — The aim of IMPACT PAD is to examine the safety and feasibility of intraprocedural flow, pressure and resistance rate changes to help predict the success of a peripheral endovascular intervention.

SUMMARY:
Defining the role of intraprocedural physiology measurements in peripheral endovascular treatment

DETAILED DESCRIPTION:
Endovascular treatment for peripheral arterial disease is commonly performed for claudication or critical limb threatening ischaemia (ischaemic rest pain, foot ulcer or gangrene). Disease is generally identified using Ankle Brachial Pressure Index or Toe Brachial Pressure Index and then lesions delineated using Doppler ultrasound or CT angiography. Clinical severity is staged using absolute walking distance (metres) in claudicants or the Society for Vascular Surgery wIfI (wound, ischaemia, foot infection) score in critical limb threatening ischaemia patients.

Intra-procedural lesion assessment and quality control is currently performed anatomically using angiography alone, with a few centres using pullback pressures across a lesion to give supplementary trans-lesional gradients or intravascular ultrasound (IVUS) to give pre and post intervention diameter and vessel area measurements. No direct or quantitative assessment of flow, or pressure normalisation across lesions is currently performed during interventions to improve blood flow to the leg.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Peripheral arterial stenosis scheduled for endovascular treatment

Exclusion Criteria:

* < 18 year of age
* Unable to give informed consent
* Estimated GFR ≤30 mL/min
* Dialysis dependent
* Unable to receive antiplatelets or periprocedural anticoagulation
* Pregnancy or breastfeeding
* Contraindication to adenosine (severe asthma or COPD)
* WIfI ulcer score <2 (no exposed bone)
* WIfI infection score <2 (skin and subcutaneous tissues only)
* WIfI gangrene score <3 (limited to digits)
* COVID-19 positive
* NYHA IV heart failure
* Contra-indication to adenosine including arrhythmia, asthma or allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-18 (Actual); Primary Completion 2024-10-06 (Estimated); Study Completion 2024-10-06 (Estimated)

PRIMARY OUTCOMES:
Pressure wire measurements | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ankur Thapar, MBBS, Principal Investigator — Mid and South Essex NHS Foundation Trust
Locations (1):
- Essex Cardiothoracic Centre, Basildon, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No